CLINICAL TRIAL: NCT00936832
Title: Front-line Combination Therapy of Sunitinib Malate Plus Chemotherapy With Leucovorin/5-Fluorouracil and Irinotecan (FOLFIRI) for Rectal Cancer Patients With Synchronous Non-Resectable Metastases: A Phase II Non Controlled Study. (SUREMETS)
Brief Title: Sunitinib Malate and Combination Chemotherapy as Front-Line Therapy in Treating Patients With Metastatic Rectal Cancer That Cannot Be Removed by Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: because the sunitinib showed futility in anotehr trial
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000637832; FFCD-0801; EUDRACT-2008-005959-19; EU-20918
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2009-07

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV rectal cancer; adenocarcinoma of the rectum; liver metastases; lung metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Rectal Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin; Sunitinib; Pharmacogenomic Testing

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Drug: sunitinib malate
Other: laboratory biomarker analysis
Other: pharmacogenomic studies
Other: pharmacological study

SUMMARY:
RATIONALE: Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as irinotecan hydrochloride, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) together with sunitinib malate may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving sunitinib malate together with combination chemotherapy works as front-line therapy in treating patients with metastatic rectal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluation of the efficacy of front-line treatment with sunitinib malate and FOLFIRI chemotherapy at 3 months in patients with rectal cancer and synchronous metastases deemed unresectable in a multidisciplinary consultation.

Secondary

* Evaluate the rate of resection of secondary metastases and rectal cancer, rate of R0 resection of metastases and rectal cancer, and the rate of complete response after resection.
* Evaluate the rate of local failure (progression of rectal cancer).
* Evaluate the rate of local complications.
* Evaluate disease-free survival.
* Evaluate progression-free survival, metastatic progression-free survival, and local progression-free survival.
* Evaluate symptom-free survival.
* Evaluate overall survival.
* Evaluate quality of life, specifically fatigue and global health score (EORTC QLQ-C30).
* Evaluate the tolerance to treatment.
* Conduct translational research, in particular, pharmacokinetic studies of plasma and rectal tumor biopsies, and histological and molecular studies.

OUTLINE: Patients receive simplified FOLFIRI chemotherapy comprising irinotecan hydrochloride IV over 90 minutes, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46 hours on days 1, 15, and 29. Patients also receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

Patients may undergo surgical resection and/or local radiotherapy if the tumor regresses. After resection or radiotherapy, patients may undergo up to 4 more courses of study treatment.

Biopsies of the tumor and healthy mucosa are collected for translational research at baseline. Blood samples are collected for pharmacodynamic and pharmacogenetic studies at baseline and at week 6. Patients also complete a quality-of-life questionnaire (EORTC QLQ-C30) at baseline and periodically thereafter.

After completion of study therapy, patients are followed up every 12 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the rectum

  * Lower pole of the tumor < 12 cm from the anal margin
* Synchronous metastases of the liver and/or lung

  * Unresectable or resectability uncertain according to the decision of a local multidisciplinary consultation
* Lesions measurable in 1 dimension by RECIST criteria (metastases and primary rectal cancer)
* No rectal obstruction requiring surgery or the emergency fitting of a prosthesis
* No CNS metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine clearance ≥ 60 mL/min
* Hemoglobin ≥ 10 g/dL (transfusions allowed)
* FEV ≥ 50%
* QT interval ≤ 450 ms (in men) or ≤ 470 ms (in women)
* Total bilirubin ≤ 1.5 times upper limit of normal
* Serum albumin ≥ 25 g/L
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No history of another cancer except for nonmelanoma skin cancer or curatively treated carcinoma in situ of the cervix

  * History of other cancers allowed provided the patient has been disease-free > 3 years
* None of the following:

  * Congestive heart failure or coronary heart disease
  * Myocardial infarction within the past year
  * Uncontrolled hypertension (systolic BP > 160 mm Hg or diastolic BP > 100 mm Hg) despite optimal medical management
* No active severe rectal bleeding
* No liver failure
* No known Gilbert syndrome
* No severe uncontrolled infection
* No chronic diarrhea, malabsorption syndrome, or intestinal obstruction/subocclusion
* No severe uncontrolled pain (visual analogue scale 5/10) with morphine treatment
* No other medical, psychological, or social condition that, in the investigator's opinion, could affect the patient's compliance with study treatment
* No hypersensitivity to any component of study treatment

PRIOR CONCURRENT THERAPY:

* See Patient Characteristics
* No prior radiotherapy to the pelvis
* More than 4 weeks since prior experimental therapy
* More than 7 days since prior CYP3A4 inhibitor before the administration of sunitinib malate
* More than 12 days since prior CYP3A4 inducer
* No concurrent participation in another clinical study
* No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03-24 (Actual); Study Completion 2010-03-24 (Actual)

PRIMARY OUTCOMES:
Response rate at 3 months as assessed by RECIST criteria

SECONDARY OUTCOMES:
Rate of complete response after resection
Rate of R0 resection of metastases
Rate of local failure
Rate of local complications
Metastatic progression-free survival
Local progression-free survival
Disease-free survival
Symptom-free survival
Overall survival
Quality of life, specifically fatigue and global health score (EORTC QLQ-C30)
Time to deterioration of the final score for overall health and fatigue
Tolerance and incidence of side effects as assessed by NCI CTCAE v2
Translational research including pharmacodynamic studies of plasma and rectal tumor biopsies and histological and molecular studies

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Rougier, MD, Principal Investigator — Hopital Ambroise Pare
Locations (1):
- Hopital Ambroise Pare, Boulogne-Billancourt, France